CLINICAL TRIAL: NCT01228825
Title: Evaluation of Plasma Concentrations and Pharmacokinetics of Cefuroxime Administered Prophylactically in Patients Undergoing Coronary Surgery With Cardiopulmonary Bypass
Brief Title: Pharmacokinetics of Cefuroxime in Cardiac Surgery With Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Santa Genoveva Hospital, Goiania GO, Brazil (Unknown)
Responsible Party: Maria José Carvalho Carmona, University of Sao Paulo
Other Study IDs: SDC2760/06/005
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Cardiopulmonary bypass; Antibiotic prophylaxis; Cefuroxime

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected sequentially after the administration of initial bolus of cefuroxime every 15 minutes during the first hour, then within two, three and six hours.
  Samples were also collected every 15 minutes during CPB. Group Off-Pump had equivalent collections, considering the time after heparinization and anastomosis initiation. Four other blood samples were collected at times considered as high risk for bacterial contamination, i.e.
  chest incision, beginning of anastomosis, after protamine administration, and chest suture.
  After each bolus of 750 mg, samples were collected within 30 minutes, one, three, and six hours.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CABG without CPB: Patients undergoing coronary artery bypass graft (CABG) without Cardiopulmonary bypass ( CPB)
- CABG with CPB: Patients undergoing coronary artery bypass graft (CABG) with cardiopulmonary bypass (CPB)

SUMMARY:
Infection, especially mediastinitis, is major complication in cardiac surgery. Considering that cardiopulmonary bypass (CPB) can alter kinetics of drugs, including antibiotics, the aim of this study was to evaluate the influence of cardiopulmonary bypass ( CPB) on plasma concentrations and pharmacokinetics of cefuroxime, administered prophylactically, in a 1.5g dose, followed by three bolus of 750mg every 6 hours, for 24 hours, in 19 patients undergoing coronary artery bypass graft (CABG) with CPB (CPB Group, n = 10), or without CPB (Off-Pump Group, n = 9); and assess whether the proposed dosing regimen is adequate to maintain plasma concentrations above 16 g/L (4 times the MIC) for the first 24 hours after the beginning of surgery.

DETAILED DESCRIPTION:
In cardiac surgery, the use of cardiopulmonary bypass may alter the kinetics and plasma concentration of drugs, including antibiotics. On the other hand, infection of the surgical field and/or mediastinitis are serious complications of cardiac surgery, with incidence ranging from 1.9 to 15%, especially when considering the lower limb infections. Inadequate prophylactic antibiotic therapy, besides not preventing infection, it can select resistant microorganisms. The second-generation of cephalosporin antibiotics have been the most used as prophylactic antibiotic for cardiac surgery due to its low toxicity and cost, good tissue penetration, good spectrum of activity against bacterias that often cause postoperative infection, i.e. Staphylococcus aureus and coagulase negative Staphylococcus, which colonize the patients' skin, and Escherichia coli, Klebsiella spp, Enterobacter spp, Proteus spp, and Pseudomonas spp, bacteria common in the lower limb or perineum which may contaminate the chest or the location of the saphenectomy. Regarding cefuroxime, it is important that the plasma concentration four times higher than the MIC (minimal inhibitory concentration), i.e. 16 g/L is maintained throughout the surgical procedure.

However, there is no consensus on the ideal dosage to be used to maintain this concentration for prevention of infection in patients undergoing cardiac surgery with cardiopulmonary bypass (CPB). Nascimento et al. demonstrated that, in patients undergoing coronary artery bypass graft (CABG) with CPB, the cefuroxime in a dose of 1.5 g every 12 hours, for 24 hours showed plasma concentrations below antibiotic prophylaxis with 16 g/L MIC after the ninth hour.

After these results, the institutional dosing changed to 1.5 g bolus at induction of anaesthesia, followed by a bolus of 750 mg every 6 hours, for 24 hours. It is necessary a study to test this dosing regimen and the influence of CPB on plasma concentrations and pharmacokinetics of cefuroxime

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for coronary surgery

Exclusion Criteria:

* Patients over 75 years old,
* body mass index (BMI) over 35 kg/m2,
* left ventricle ejection fraction below 35%,
* serum creatinine greater than or equal to 1.4 mg/dL,
* prothrombin activity lower than 80%,
* serology positive for hepatitis,
* use of oral anticoagulants,
* allergy to cefuroxime

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients scheduled for coronary surgery were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the influence of CPB on plasma concentrations and pharmacokinetics of cefuroxime | 24 hours
  Some authors argue that CPB could trigger a drop in the drug plasma concentration due to hemodilution, changes in volume of distribution, redistribution of blood flow to peripheral tissue, vasodilatation due to inflammatory, drug sequestration by the CPB circuit and/or the lungs. Others argue the pharmacokinetics of water-soluble cephalosporin showed that the rate of elimination is dependent on renal function, with reduction of plasma clearance, prolongation of biological half-life, and elevated plasma concentrations at the end of CPB.

SECONDARY OUTCOMES:
Assess whether the proposed dosing regimen is adequate to maintain plasmaconcentrations above (4 times the MIC). | 24 hours
  Nascimento et al. (2005) demonstrated that, in patients undergoing coronary artery bypass graft (CABG) with CPB, antibiotic prophylaxis with cefuroxime in a dose of 1.5 g every 12 hours, for 24 hours showed plasma concentrations below MIC (16 g/L) after the ninth hour. After these results, the institutional dosing changed to 1.5 g bolus at induction of anaesthesia, followed by a bolus of 750 mg every 6 hours, for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana AP Bosco Ferreira, MD, Principal Investigator — University of Sao Paulo; Maria Jose C Carmona, phD, Study Chair — University of Sao Paulo
Locations (1):
- Heart Institute University of Sao Paulo, São Paulo, São Paulo, Brazil